CLINICAL TRIAL: NCT01031966
Title: A Pilot, Randomized, Open-label Study in Patients on Chronic Dialysis With End Stage Renal Disease (Esrd), to Evaluate the Enhancing Effect of Two Doses of Thymosin Alpha 1 on the Immunogenicity of h1n1sw Monovalent Vaccine
Brief Title: A Pilot Study to Evaluate ZADAXIN's® (Thymalfasin) Ability to Enhance Immune Response to the H1N1sw Influenza Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: sigma-tau i.f.r. S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ST1472-DM-09-005
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: END STAGE RENAL DISEASE
Keywords: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — focetria; Thymalfasin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- H1N1sw monovalent vaccine (Active Comparator)
  Interventions: Biological: MF59 adjuvanted H1N1 influenza monovalent vaccine
- Thymosin alpha 1 3.2mg (Experimental)
  Interventions: Drug: Thymosin alpha 1
- Thymosin alpha 1 6.4 mg (Experimental)
  Interventions: Drug: Thymosin alpha 1

INTERVENTIONS:
Biological: MF59 adjuvanted H1N1 influenza monovalent vaccine — One/two single administration
  Other Names: Focetria™
  Arms: H1N1sw monovalent vaccine
Drug: Thymosin alpha 1 — 1.6 mg, 3.2 mg seven days before vaccination (study day -7) and at the same day of vaccination (study day 0)
  Other Names: Zadaxin
  Arms: Thymosin alpha 1 3.2mg
Drug: Thymosin alpha 1 — 1.6 mg, 6.4 mg seven days before vaccination (study day -7) and at the same day of vaccination (study day 0)
  Other Names: Zadaxin
  Arms: Thymosin alpha 1 6.4 mg

SUMMARY:
The purpose of this explorative trial is to collect preliminary data on efficacy and safety of thymosin alpha 1 given at different doses as an adjuvant to egg-derived H1N1sw monovalent influenza vaccine in hemodialysis patients. The final aim is that of gathering information needed for planning a following confirmatory study on the efficacy and safety of Thymosin alpha 1 in the same indication.

DETAILED DESCRIPTION:
The emergence and spread of the novel influenza A (H1N1) virus has been of great concern globally.

Uremic patients are especially vulnerable to infections and it is generally recommended to vaccinate patients with chronic renal insufficiency yearly against influenza. In patients on haemodialysis (HD) the vaccination response has been considered suboptimal.

Decreased antibody response to T-cell dependent antigens may be one factor that accounts for insufficient efficacy of certain vaccination programs (eg, influenza). Diminished antibody responses have also been reported in patients with end-stage renal disease. The evidence for impairment of cell-mediated immunity in hemodialysis patients has been attributed to incompetence in T-cell-mediated immune responses.

Since Zadaxin can enhance T-cell-dependent specific antibody production, the addition of Zadaxin (Thymosin alpha 1)to vaccination programs for immunocompromised individuals should be effective.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Age > 18 .
3. Chronic dialysis for ESRD .
4. Life expectancy of at least 6 months.

Exclusion Criteria:

1. They have any serious disease
2. They are hypersensitive to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the vaccine.
3. They have a history of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine.
4. Within the past 3 days, they have experienced fever (i.e., axillary temperature _ 38°C).
5. They have any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objective.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The measures of immunogenicity, as determined by HI; MN and SRH | Geometric mean HI titer (GMT) on Day 0, Day 21, Day 42, Day 84 and Day 168 for the primary course

CONTACTS AND LOCATIONS:
Overall Officials: Agostino Naso, MD, Principal Investigator — Second Division of Nephrology and Dialysis - Padua Hospital
Locations (1):
- Second Division of Nephrology and Dialysis - Padua Hospital, Padua, Italy